CLINICAL TRIAL: NCT06294067
Title: A Double Blinded Randomized Control Trial to Aid in Determining the Dose Dependent Relationship of Docosahexaenoic Acid (DHA) on Eicosapentaenoic Acid (EPA) Feedback Inhibition Using Carbon 13 as a Biomarker
Brief Title: A Dose Response Investigation of Docosahexaenoic Acid (DHA)
Acronym: DRI-DHA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Richard Bazinet, Principle Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 43261
Record Dates: First submitted 2023-09-25; First posted 2024-03-05 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Nutrition, Healthy
Keywords: docosahexaenoic acid; eicosapentaenoic acid; dietary reference intakes; retroconversion
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: Double blinded, randomized, control, dose-response supplementation trial
Who Masked: Participant, Investigator
Masking Description: Block Randomization was used to ensure that sample sizes remain balanced throughout the study. Following successful completion of informed consent, the questionnaire and anthropometric assessment participants will be randomized into groups, of a possible six, using a blocked (Latin squares) randomization. These groups will represent DHA0 (0mg/d), DHA1 (100mg/d), DHA2 (200mg/d), DHA3 (400mg/d), DHA4 (800mg/d), and DHA5 (1000mg/d) groups. The Latin square sequences will be randomly allocated to participants with a similar number of participants allocated to each treatment sequence. The participants will only be randomized once all information is collected, informed consent has been obtained and questionnaires have been filled out following the first study call/zoom meeting. Then following their first study in person visit and post blood sample extraction they will be given their DHA capsules, which have been organized by a lab member not directly involved in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- DHA0 - 0mg of DHA/d (Placebo Comparator): DHA0 participants are in the placebo group and will take 5 soybean oil based capsules per day and will not receive any DHA. Every group takes 5 capsules per day to maintain blinding.
  Interventions: Dietary Supplement: soybean oil placebo
- DHA1 - 100mg of DHA/d (Active Comparator): DHA1 participants will take 100mg/d of DHA. As the DHA supplements are 200mg of DHA per capsule the participants here will take one 200mg capsule every other day and the rest of the capsules will be placebos.
  Interventions: Dietary Supplement: docosahexaenoic acid (DHA)
- DHA2 - 200mg of DHA/d (Active Comparator): DHA2 participants will take one 200mg capsule of DHA and 4 placebos per day.
  Interventions: Dietary Supplement: docosahexaenoic acid (DHA)
- DHA3 - 400mg of DHA/d (Active Comparator): DHA3 participants will take two 200mg capsules of DHA and 3 placebos per day.
  Interventions: Dietary Supplement: docosahexaenoic acid (DHA)
- DHA4 - 800mg of DHA/d (Active Comparator): DHA4 participants will take four 200mg capsules of DHA and 1 placebo per day.
  Interventions: Dietary Supplement: docosahexaenoic acid (DHA)
- DHA5 - 1000mg of DHA/d (Active Comparator): DHA5 participants will take five 200mg capsules of DHA and no placebos per day.
  Interventions: Dietary Supplement: docosahexaenoic acid (DHA)

INTERVENTIONS:
Dietary Supplement: docosahexaenoic acid (DHA) — 72 healthy participants will be divided into 6 groups and receive varying amounts of DHA (0mg, 100mg, 200mg, 400mg, 800mg and 1000mg) over the course of 8 weeks.
  Arms: DHA1 - 100mg of DHA/d; DHA2 - 200mg of DHA/d; DHA3 - 400mg of DHA/d; DHA4 - 800mg of DHA/d; DHA5 - 1000mg of DHA/d
Dietary Supplement: soybean oil placebo — 72 healthy participants will be divided into 6 groups and receive varying amounts of DHA (0mg, 100mg, 200mg, 400mg, 800mg and 1000mg) over the course of 8 weeks. The 0mg group will receive only placebos.
  Arms: DHA0 - 0mg of DHA/d

SUMMARY:
Docosahexaenoic acid (DHA) is an omega-3 polyunsaturated fatty acid (n-3 PUFA), commonly consumed from fish, that regulates many critical functions within the body including the brain, eye, and heart. While the metabolic precursor to DHA, alpha-linolenic acid (ALA) is considered nutritionally essential and has a set Dietary Reference Intake (DRI), DHA has not yet been deemed essential and does not have a set DRI. Currently, research suggests an intake range of dietary DHA to be anywhere from 0 to over 500mg/d. The aim of our study is to further investigate a feedback mechanism or accumulation that occurs with eicosapentaenoic acid (EPA) as a result of increased dietary DHA to provide insight for potential Recommended Dietary Intake (RDI) values.

Hypothesis: The dietary DHA dose at which blood EPA levels increase is the point at which elongation slows, indicating a significant negative feedback pathway is present.

Objectives: 1: To determine the dose-response for DHA to increase blood EPA levels in a mixed vegetarian and vegan population. 2: Investigate the DHA dose and time at dose that increases EPA using natural abundance delta carbon-13 (δ13C) as a tracer. 3: To measure DHA turnover and loss rates. 4: Provide data for exploratory analyses related to PUFA metabolism and the effect of DHA on disease related biomarkers.

Method: During an 8-week trial, 72 healthy vegan or vegetarian males and females (18-50 years) will be supplemented with 1 of 6 algal-oil based DHA doses: 0, 100, 200, 400, 800 or 1000 mg/d. Blood will be collected at days 0, 3, 7, 14, 28 and 56 and will be analyzed for changes in blood EPA levels as the primary outcome and plasma δ13C EPA signature as the secondary outcome.

Significance: Investigating this negative feedback pathway is of great importance in providing evidence to support n-3 PUFA DRIs. EPA and DHA are ecologically sensitive with their major source coming from unsustainably farmed fish stocks and having a set DRI may help to limit the overconsumption of these nutrients.

DETAILED DESCRIPTION:
Docosahexaenoic acid (DHA) is vital for the structure of cell membranes, essential for brain and eye development, found at high levels throughout the brain and nervous system and is important for optimal cognitive development in children, the growth of the fetus during pregnancy and healthy breast milk during lactation. DHA has also been shown to aid in the protection against primary and secondary symptoms of cardiovascular disease as well as macular degeneration. However, whether DHA is deemed to be essential in the diet remains controversial. Meanwhile, the Institute of Medicine (now the National Academy of Medicine) set an adequate intake for DHA's precursor, alpha-linolenic acid (ALA), at 1.6 g/d and 1.1 g/d for healthy males and females, respectively. The investigators believe the confusion arises from the approach to studying omega-3 fatty acids, particularly DHA requirements. For these studies, DHA is supplemented, and often complex, multifactorial disease outcomes are used as endpoints. The doses of DHA used in these studies are often subjective and participants, including controls, have varying DHA intakes and levels. Supplementing a population, like vegetarians or vegans whose levels are similarly low would be useful. Classically, it was believed that that when DHA is consumed a portion is converted "backwards" to eicosapentaenoic acid (EPA) which then accumulates in a process called "retroconversion." However, using a novel approach called compound-specific isotope analysis (CSIA), the investigators observed that the rise in EPA is not primarily from retroconversion, but rather from a backlog of EPA primarily originating from ALA. Initially demonstrated in rodent models by CSIA, the team confirmed by similar modeling that DHA consumption in humans results in the same backlog of EPA. Critically, DHA induces a backlog in metabolism of EPA and dietary ALA appears to be essential for this backlog. Thus, the increase in EPA represents a biochemical feedback pathway that slows DHA synthesis in response to sufficient DHA.

Significance: By precisely determining the lowest amount of DHA required to activate this feedback mechanism it may be useful for future estimation of DHA requirements. Moreover, the problem with the amounts suggested for the unofficial recommendations is that if the global population were to consume these amounts it would be environmentally concerning as this nutrient is ecologically sensitive with its major source coming from already stressed ocean fish stocks, encouraging unsustainable fishing practices, something environmentalists and researchers have said are creating legitimate climate and health concerns.

Hypothesis: The dose at which EPA increases with increased DHA is the point at which elongation slows, indicating a significant feedback pathway is present.

Objectives: 1. To determine the dose-response for DHA to increase EPA. 2. Investigate the DHA dose and time that increases EPA using CSIA. 3. To measure EPA, DPAn-3, and DHA turnover and loss rates. 4. Provide data for exploratory analysis related to PUFA metabolism, ALA consumption and its effect on EPA and DHA levels, and DHA's effects on disease related biomarkers, C-Reactive Protein (CRP), and blood clotting.

Trial Design: Co-principle investigators Dr. Richard Bazinet and Dr. John Sievenpiper and co-investigators, Drs. David Jenkins and Adam Metherel along with PhD student Amy Symington, will conduct a double blinded, placebo-controlled, dose-response supplementation trial. Seventy-two healthy vegans or vegetarians who are 18-50 years old will be randomly assigned to 1 of 6 groups. Prior to randomization, participants will undergo a 2-week run-in phase to gather their questionnaire data. Once randomized, each group will take DHA supplements of either 0mg (placebo), 100mg, 200mg, 400mg, 800mg and 1000mg per day over the course of 8 weeks. These doses represent the range of DHA intake levels spanning average population intakes (<100 mg/d), frequently recommended intakes (250 - 500 mg/d), and DHA intake levels known to increase plasma EPA levels (1000 mg/d). A questionnaire will be administered to obtain information in relation to approximate ALA, EPA and DHA intake before and after the supplementation period. A 3-day weighed diet diary will be provided to obtain food intake over the course of the supplementation period to gauge ALA consumption. Participants will be asked to refrain from DHA rich foods during the supplementation period. This will not be an issue as this population generally do not consume DHA rich foods. Baseline intake of the essential fatty acid ALA will be assessed via questionnaire and verified by blood samples.

Participants: The study will recruit 72 healthy vegetarians and vegans to allow for the lowest possible baseline EPA and DHA levels. Exclusion criteria are as follows: consumption of EPA and/or DHA supplement within the past six months, have 3% or higher of DHA in their total plasma lipids, BMI <18 kg/m2 or >30 kg/m2, are menopausal or post-menopausal, pregnant or breastfeeding, chronic or communicable diseases (like multiple sclerosis, kidney and inflammatory bowel disease, Type 2 diabetes, cancer or heart disease), use of chronic anti-inflammatory medication, use of lipid-controlling medication, hypertriglyceridemia (>4 mmol/l) or hypercholesterolemia (LDL-C >5 mmol/l), anticipate major changes in lifestyle, smoker, heavy alcohol user (>3 drinks/day) and major surgery or has participated in an intervention trial in the last six months. This exclusion data is in line with previous meta-analyses and n-3 supplementation trials that have used the above exclusion criteria as they affect n-3 PUFA metabolism. Participants who sign the consent form who are later deemed to be ineligible due to BMI or % of DHA levels will be informed via email and/or phone. This is explained in the consent form.

Fatty acid analyses: Blood samples for baseline and follow-up meetings will be obtained following an overnight 12-hour fast. Blood samples will be collected at days 0, 3, 7, 14, 28 and 56. The samples will be collected by a registered nurse. Whole blood samples will be saved and stored from each participant. Then, the remaining whole blood samples from each participant will be centrifuged and the plasma and red blood cells (RBCs) isolated from each sample. They will be stored at -80°C in an air tight container until required for analysis. Plasma and RBCs samples will be analyzed for fatty acid concentrations using gas chromatography (GC)-flame ionization detection and delta carbon-13 (δ13C) will be assessed using GC-isotope ratio mass spectrometry. Plasma and RBCs will be analyzed with changes in plasma EPA levels as the primary outcome and plasma δ13C EPA signature, measured by compound specific isotope analysis (CSIA), as the secondary outcome. The δ13C signature of EPA will also be measured to see that it aligns with the δ13C signature of plasma ALA and not the DHA supplement.

Sample Size: Power was calculated based on results from the literature which has consistently reported changes in plasma EPA following DHA supplementation for 6 weeks with 12 subjects, and is consistent with our findings. Using means, standards deviations and sample sizes from the Metherel et al study in 2019 and these two previous studies, an alpha = 0.05 and desired power of 0.8 we determined sample sizes of just over 9 as sufficient to yield a statistically significant effect. As such, to account for a projected 20-25% dropout rate we will recruit 12 participants to ensure we are appropriately powered for our primary outcome.

Secondary analysis: Depending upon recruitment the investigators will examine if males and females respond differently in an exploratory analysis, recognizing they may not be powered to detect potentially real, but small sex-related differences. The investigators will use whole blood samples collected to determine FADS1, FADS2, ELOVL2 and ELOVL5 isoforms which have been shown to affect blood levels of EPA and DHA as a sub analysis.

The investigators will also provide data to do additional analysis related to n-3 PUFA turnover and loss rates, participants' ALA consumption and its effect on n-3 PUFA metabolism. In addition, some of the beneficial outcomes that may occur with DHA supplementation according to current research will be determined, including blood pressure, heart rate, triglycerides, and LDL, HDL and total cholesterol.

Recruitment: Participants will be recruited by way of email and social media to various vegetarian/vegan focused groups and organizations.

Anthropometric analyses: Height will be measured with a wall-mounted stadiometer.

Body weight will be assessed by beam scale. Waist circumference will be assessed using the Heart and Stroke Foundation methodology. Blood pressure (BP) and resting heart rate will be measured. To collect this measure, participants will remain seated in a quiet, temperature-controlled room for at least 5 minutes to achieve resting heart rate and BP. Subsequently, BP will be measured oscillometrically using the OMRON Intellisense HEM-907 according to JNC VII criteria. BP will be measured in triplicate, with each measurement separated by one minute, and the average of the three measures will be taken.

Biochemical analyses: Plasma and RBC samples for EPA and DHA will be separated by centrifuge and immediately frozen at -80 C at the University of Toronto for later analysis. Although plasma is the primary focus for the outcome, both plasma and RBC samples will be analyzed for comparison using GC-FID to determine EPA and DHA levels and δ13C will be analyzed using GC-IRMS.

Baseline and follow-up questionnaire: To obtain approximate ALA, EPA and DHA intake both before and after the supplementation period, a questionnaire will be provided to participants via email to fill out following the first phone/zoom meeting and at the final visit on day 56.

Statistical Analysis

Primary outcomes. Plasma and red blood cell (RBC) samples will be analyzed using GC-FID to determine n-3 PUFA concentrations within each group. Statistical analysis will be performed by a two-way ANOVA (dose x time) with repeated measures on time to determine interaction and/or main effects. In addition, the increase in EPA levels will be analyzed by segmented regression (or breakpoint analysis), as is done with the indicator amino acid oxidation technique between doses and within each time point to identify the dose of DHA supplementation that results in a sudden increase in EPA levels, the DHA dose that initiates feedback inhibition. Repeated measures post hoc Tukey test will be used to determine significant differences in DHA% and EPA% between visits as well as between groups. A Games-Howell test would be administered during the Tukey test if a group happens to have uneven participant numbers due to dropouts.

Secondary outcomes. δ13C will be analyzed using GC-IRMS. The δ13C signature of EPA will be measured to see that it aligns with the δ13C signature of plasma ALA and not the DHA supplement. Turnover rates and half-lives of EPA, DPAn-3 and DHA will be calculated by GraphPad Prism version 10.0 and the rate of loss of EPA, DPAn-3 and DHA in nmol/ml/day from the plasma will be calculated using the following formula: Jout = 0.693CFA/t1/2.

Exploratory and adherence outcomes. Repeated measures mixed effect models will be used to assess changes in all exploratory outcomes without controlling for false discovery rate. Pairwise comparisons between groups will be performed using Tukey-Kramer adjustment or other appropriate statistics. Effect modification by ALA consumption, sex, and genetics will be explored and blood samples will be analyzed for compliance.

Subgroup Analysis. A priori analysis will be conducted by age, sex, ethnicity, baseline BMI, baseline waist circumference, genetic variants and ALA consumption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy vegans or vegetarians who do not consume meat or fish.

Exclusion Criteria:

* Has regularly consumed EPA and/or DHA supplements within the past six months
* Having 3% or higher of DHA in their total plasma lipids
* BMI <18 kg/m2 or >30 kg/m2
* Menopausal or post-menopausal
* Pregnant or breastfeeding
* Has a chronic or communicable diseases (like multiple sclerosis, kidney and inflammatory bowel disease, Type 2 diabetes, cancer or heart disease)
* Suffers from acute or chronic infections, use of chronic anti-inflammatory medication, use of lipid-controlling medication, hypertriglyceridemia (>4 mmol/l) or hypercholesterolemia (LDL-C >5 mmol/l)
* Anticipates major changes in lifestyle
* Is a smoker
* Is a heavy alcohol user (>3 drinks/day)
* Has had a major surgery involving organs like open heart surgery or organ transplants in the last six months
* Is or has participated in an intervention trial in the last six months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Changes in omega-3 polyunsaturated fatty acid (n-3 PUFA) blood levels | 8 weeks
  Changes in blood n-3 PUFA levels within the various groups and at what day a rise in EPA occurs at.

SECONDARY OUTCOMES:
Changes in the delta carbon 13 (δ13C) n-3 PUFA signatures | 8 weeks
  Using δ13C as a tracer the change in δ13C n-3 PUFA signatures will be investigated to determine whether the EPA is coming from dietary sources or retroconversion of the DHA supplement.
Measure of n-3 LC PUFA turnover rates | 8 weeks
  From the change in n-3 LC PUFA δ13C signatures investigators will be able to determine n-3 LC PUFA turnover rates in days.
Measure of n-3 LC PUFA half-lives | 8 weeks
  From the change in n-3 LC PUFA δ13C signatures investigators will be able to determine n-3 LC PUFA half-lives or rate of loss in nmol/ml/day.

OTHER OUTCOMES:
Increased intake of dietary α-Linolenic acid (ALA) and the inhibition of long chained omega-3 polyunsaturated fatty acids (LC n-3 PUFA) synthesis | 8 weeks
  How increased dietary ALA (mg/d) during DHA supplementation inhibits or slows LC n-3 PUFA synthesis will be investigated.
Comparing the potential change in omega-3 long chained polyunsaturated fatty acids (n-3 LC PUFA) levels between male and female participants | 8 weeks
  Other research studies have shown N-3 LC PUFA synthesis to be higher in females due to an estrogen-induced increase in LC n-3 PUFA synthesis as a result of estrogen's upregulation of rate limiting enzyme, ELOVL2. The difference in LC n-3 PUFA levels, particularly DHA, between sexes will be investigated in this study.
Comparing the potential change in n-3 LC PUFA δ13C signatures between male and female participants | 8 weeks
  Other research studies have shown N-3 LC PUFA synthesis to be higher in females due to an estrogen-induced increase in LC n-3 PUFA synthesis as a result of estrogen's upregulation of rate limiting enzyme, ELOVL2. The difference in LC n-3 PUFA δ13C signatures, particularly DHA, between sexes will be investigated in this study.
Comparing the potential change in n-3 LC PUFA levels between genetic variations | 8 weeks
  Other research studies have shown genetic variation in polyunsaturated fatty acid metabolism, particularly in the fatty acid desaturase (FADS) gene cluster and fatty acid elongase (ELOVL) gene family. As a result, the investigators will look at various genes and single nucleotide polymorphisms (SNPs) that have been shown to influence synthesis through the change in n-3 LC PUFA levels in this study.
Comparing the potential change in n-3 LC PUFA δ13C signatures between genetic variations | 8 weeks
  Other research studies have shown genetic variation in polyunsaturated fatty acid metabolism, particularly in the fatty acid desaturase (FADS) gene cluster and fatty acid elongase (ELOVL) gene family. As a result, the investigators will look at various genes and single nucleotide polymorphisms (SNPs) that have been shown to influence synthesis through the change in n-3 LC PUFA δ13C signatures.
Changes in cardiovascular disease (CVD) biomarkers (BMI in kg/m^2) | 8 weeks
  Change in participants' body mass index (BMI) (kg/m^2) will be investigated as an indicator of CVD onset.
Changes in cardiovascular disease (CVD) biomarkers (Waist circumference in cm/inch) | 8 weeks
  Change in participants' waist circumference (cm/inch), will be investigated at as an indicator of CVD onset.
Changes in cardiovascular disease (CVD) biomarkers (blood pressure in mmHg) | 8 weeks
  Change in participants' blood pressure (mmHg) will be investigated at as an indicator of CVD onset.
Changes in cardiovascular disease (CVD) biomarkers (heart rate in beats per minute) | 8 weeks
  Change in participants' heart rate (beats per minute) will be investigated at as an indicator of CVD onset.
Changes in cardiovascular disease (CVD) biomarkers (blood lipid profile changes in mmol/L) | 8 weeks
  Change in participants' blood lipid profile including triglycerides, LDL, HDL, and total cholesterols (mmol/L) levels will be investigated as indicators of CVD onset.
Changes in δ13C DHA signature levels to document adherence | 8 weeks
  Adherence outcomes will be based on the participant's measured changes in δ13C DHA signature levels (per mil, ‰).

CONTACTS AND LOCATIONS:
Overall Officials: Richard P Bazinet, PhD, Principal Investigator — University of Toronto
Locations (1):
- Clinical Nutrition and Risk Factor Modification Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
None at the moment

REFERENCES:
- [Background] Li J, Pora BLR, Dong K, Hasjim J. Health benefits of docosahexaenoic acid and its bioavailability: A review. Food Sci Nutr. 2021 Jul 23;9(9):5229-5243. doi: 10.1002/fsn3.2299. eCollection 2021 Sep. PMID 34532031
- [Background] Abdelhamid AS, Brown TJ, Brainard JS, Biswas P, Thorpe GC, Moore HJ, Deane KH, Summerbell CD, Worthington HV, Song F, Hooper L. Omega-3 fatty acids for the primary and secondary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2020 Feb 29;3(3):CD003177. doi: 10.1002/14651858.CD003177.pub5. PMID 32114706
- [Background] Metherel AH, Irfan M, Klingel SL, Mutch DM, Bazinet RP. Compound-specific isotope analysis reveals no retroconversion of DHA to EPA but substantial conversion of EPA to DHA following supplementation: a randomized control trial. Am J Clin Nutr. 2019 Oct 1;110(4):823-831. doi: 10.1093/ajcn/nqz097. PMID 31204771
- [Background] Metherel AH, Chouinard-Watkins R, Trepanier MO, Lacombe RJS, Bazinet RP. Retroconversion is a minor contributor to increases in eicosapentaenoic acid following docosahexaenoic acid feeding as determined by compound specific isotope analysis in rat liver. Nutr Metab (Lond). 2017 Nov 28;14:75. doi: 10.1186/s12986-017-0230-2. eCollection 2017. PMID 29209405
- [Background] Schuchardt JP, Ostermann AI, Stork L, Kutzner L, Kohrs H, Greupner T, Hahn A, Schebb NH. Effects of docosahexaenoic acid supplementation on PUFA levels in red blood cells and plasma. Prostaglandins Leukot Essent Fatty Acids. 2016 Dec;115:12-23. doi: 10.1016/j.plefa.2016.10.005. Epub 2016 Oct 12. PMID 27914509
- [Background] Sanders TA. DHA status of vegetarians. Prostaglandins Leukot Essent Fatty Acids. 2009 Aug-Sep;81(2-3):137-41. doi: 10.1016/j.plefa.2009.05.013. Epub 2009 Jun 4. PMID 19500961
- [Background] Jenkins DJ, Sievenpiper JL, Pauly D, Sumaila UR, Kendall CW, Mowat FM. Are dietary recommendations for the use of fish oils sustainable? CMAJ. 2009 Mar 17;180(6):633-7. doi: 10.1503/cmaj.081274. No abstract available. PMID 19289808